CLINICAL TRIAL: NCT01800812
Title: Phase One Study With Direct Individual Benefit: Effects of OM-174 in Adult Patients With Solid Tumors.
Brief Title: Effects of OM-174 in Adult Patients With Solid Tumors
Acronym: OM-174
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None
Other Study IDs: BARDOU PHRC R 2002
Record Dates: First submitted 2013-02-22; First posted 2013-02-28 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Solid Tumors

INTERVENTIONS:
Biological: Injections of OM-174

SUMMARY:
Methods Patients received OM-174 twice weekly for a total of 5, 10 or 15 injections of either 600, 800 or 1000 µg/m². Pharmacokinetic analysis and cytokine dosages were performed. Natural Killer cells activity and toll-like receptors 4 polymorphism analysis were also performed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a histologically proven solid tumor, refractory to conventional treatment or for which no such treatment existed.
* At least one month since the last chemotherapy
* Life expectancy above 3 months
* Written informed consent
* Age above 18

Exclusion Criteria:

* Patient's refusal
* Infection
* Brain metastasis
* Autoimmune disease
* Regular use of steroids
* Patient included in another protocol
* Chemotherapy or radiotherapy less than 6 weeks ago
* Immunotherapy less than 8 weeks ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27
Dates: Start 2007-03; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
The occurrence of any adverse event | up to 8 weeks

REFERENCES:
- [Derived] Isambert N, Fumoleau P, Paul C, Ferrand C, Zanetta S, Bauer J, Ragot K, Lizard G, Jeannin JF, Bardou M. Phase I study of OM-174, a lipid A analogue, with assessment of immunological response, in patients with refractory solid tumors. BMC Cancer. 2013 Apr 2;13:172. doi: 10.1186/1471-2407-13-172. PMID 23547558